CLINICAL TRIAL: NCT03818191
Title: Pharmacogenomics and Pharmacometabolomics of Acamprosate Treatment Outcome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Victor M. Karpyak, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-006428; 1R01AA027486-01 (NIH); 1U01AA027487 (NIH)
Record Dates: First submitted 2019-01-14; First posted 2019-01-28 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Acamprosate (Active Comparator): All participants will be randomized to receive acamprosate or placebo in a double-blinded placebo-controlled trial.
  The most common side effect associated with acamprosate use is diarrhea, which occurs in approximately 16% of patients. Other frequently occurring side effects include asthenia, nausea, pruritus, and flatulence, headache, abdominal pain, flu syndrome, edema, weight gain, and myalgia.
  Interventions: Drug: Acamprosate
- Placebo (Placebo Comparator): All participants will be randomized to receive acamprosate or placebo in a double-blinded placebo-controlled trial.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acamprosate — The research pharmacy contracted for this study will randomize the study participants for all sites with placebo or acamprosate.
  Arms: Acamprosate
Other: Placebo — The research pharmacy contracted for this study will randomize the study participants for all sites with placebo or acamprosate.
  Arms: Placebo

SUMMARY:
AUDs are difficult to treat, and relapse rates are high, with an estimated 80% of individuals with AUDs returning to alcohol use after completing addictions treatment. Novel treatment approaches are needed to enhance long term sobriety. The investigator's research team has been investigating the use of acamprosate to prevent relapse to alcohol use. Unfortunately despite being FDA approved and endorsed by the American Psychiatric Association only 10% of patients treated for AUD are prescribed acamprosate or other antidipsotropic medications. The number is higher for patients treated in programs affiliated with Mayo Clinic Addiction Services (approximately 20%) but is way less than expected. The most common reasons behind these low numbers are the understanding that not every patient benefits from the use of specific medication and the lack of biomarkers predictive of response. The purpose of this project is to identify such biomarkers by discovery of genomic and metabolomic markers associated with response to acamprosate treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to85; DSM-5 diagnosis of AUD determined by PRISM;
2. Completion of alcohol detoxification (CIWA score < 5) and no alcohol for at least 7 days (but no more than 35 days);
3. Ability to provide informed consent
4. Ability to speak English
5. Willingness to use the study medications for 3 months and attend follow-up visits.
6. No chronic/daily use of benzodiazepines, opioids, or stimulants for a period of time which is determined by 3 x the medication half-life value (see addendum A) to be completed before the initiation of study medication (acamprosate or placebo).
7. Willingness to discontinue previously prescribed acamprosate for a period of at least 3 days before randomization to study medication (acamprosate or placebo).

Exclusion Criteria:

1. Hypersensitivity or allergy to acamprosate
2. Current use of wellbutrin and not willing to switch to an acceptable antidepressant medication
3. Renal impairment (creatinine level >1.5 mg/dL);
4. Diagnosis of advanced liver disease indicated in the medical record or by a MELD score of above 10;
5. Women who are pregnant, breastfeeding, or planning to become pregnant during the next year;
6. Primary diagnosis of substance use disorder other than alcohol as determined by PRISM or in medical record review or secondary diagnosis of active (within the past year) benzo/sedative dependence, opioid dependence, stimulant dependence, heroin dependence, and/or cocaine dependence
7. Refusal to abstain from any chronic/daily use of prescribed benzodiazepines, opioids, stimulants, cannabis related medication such as CBD or medical marijuana, during the course of participation.
8. Current use of Naltrexone and not willing to stop and switch to Acamprosate/Placebo
9. Current use of Antabuse.
10. Active suicidal ideation or any unstable medical or psychiatric condition as determined by responses to PRISM or by the investigator.
11. Status of involuntary or court-ordered admission at time of consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-11-04 (Actual); Study Completion 2023-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor M Karpyak, MD, Ph.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Hazelden Betty Ford Foundation, Center City, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Hazelden Betty Ford Foundation, Newberg, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the study began in June of 2019 and continued to July 2023 with follow-up visits completed in October 2023. All participants were recruited while attending a residential intensive treatment program.
Pre-assignment Details: Participants were evaluated by PRISM to confirm alcohol use disorder diagnosis and no secondary diagnosis of active other substance use disorder was present. Additional testing was done for renal impairment and advanced liver disease. Participants were required to be willing to stop chronic/daily use of prescribed benzodiazepines, opioids, stimulants, cannabis related medication such as CBD or medical marijuana during participation. Review of medications including anti-depressants was done.
Groups:
- Acamprosate: All participants will be randomized to receive acamprosate or placebo in a double-blinded placebo-controlled trial.
  The most common side effect associated with acamprosate use is diarrhea, which occurs in approximately 16% of patients. Other frequently occurring side effects include asthenia, nausea, pruritus, and flatulence, headache, abdominal pain, flu syndrome, edema, weight gain, and myalgia.
  Acamprosate: The research pharmacy contracted for this study will randomize the study participants for all sites with placebo or acamprosate.
Period: Overall Study
Arm/Group | Acamprosate | Placebo
Started | 184 | 104
Completed | 81 | 51
Not Completed | 103 | 53

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acamprosate | Placebo | Total
Number analyzed (Participants) | 184 | 104 | 288
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 176 | 104 | 280
  >=65 years | 8 | 0 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.986 (11.761) | 44.023 (11.071) | 45.277 (11.536)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 30 | 85
  Male | 129 | 74 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 168 | 96 | 264
  Unknown or Not Reported | 16 | 6 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 2 | 2 | 4
  White | 161 | 95 | 256
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 16 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Continuous Sobriety According to Alcohol Timeline Follow Back
Description: The Alcohol Timeline Follow Back (TLFB) is a drinking assessment method that obtains estimates of daily drinking and has been evaluated with clinical and nonclinical populations. Using a calendar, people provide retrospective estimates of their daily drinking over a specified time period that can vary up to 12 months from the interview date.
Time Frame: Will be defined as continuous sobriety (yes/no) during 3 months of treatment
Population: The analyzed sample included participants that completed 3 months of the study, as well as, those that dropped out but were known to have relapsed before 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 101 | 55
Participants | 66 | 39

2. Secondary Outcome: Day Until First Alcohol Use (Relapse) - Alcohol Timeline Follow Back
Description: as for outcome 1
Time Frame: The number of days until first alcohol use (relapse) assessed by TLFB during 3 months of treatment
Measure: Median (Inter-Quartile Range); unit: Number of days
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 127 | 70
Number of days | 80 [31.5 to 89] | 82 [43 to 89]

3. Secondary Outcome: Days Until First Relapse (Heavy Relapse) - Timeline Follow Back
Description: as for outcome 1
Time Frame: Number of days until first relapse (heavy relapse) between medication start and 3 months follow-up
Measure: Median (Inter-Quartile Range); unit: Number of days
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 127 | 70
Number of days | 81 [33 to 89] | 82.5 [52.25 to 89]

4. Secondary Outcome: Cumulative Abstinence Duration - Timeline Follow Back
Description: as for outcome 1
Time Frame: Cumulative abstinence duration proportion: proportion of days over the length of 3 month follow-up during which participants were abstinent from alcohol use, a score range of 0 (drinking continuously) to 100 (maintain complete abstinence) is applied.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 101 | 54
percentage of days | 96.57 (6.85) | 96.01 (13.90)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 3 months during each patient's participation.
Arm/Group | Acamprosate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/184 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/184 | 0/104
Other Adverse Events (participants affected / at risk) | 55/184 | 35/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acamprosate (N=184) | Placebo (N=104)
ER/Hospital visit for suicidal ideation, intoxication, or alcohol withdrawal (Psychiatric disorders) | 7 (8) | 3 (3)
Loss of sexual interest or problems with erection or achieving orgasm (Reproductive system and breast disorders) | 4 (4) | 3 (3)
Prolonged QT interval (Cardiac disorders) | 0 (0) | 1 (1)
Headache/Migraine (Nervous system disorders) | 5 (5) | 2 (2)
Cold/Flu (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (5)
Jaw and Ear Pain, Broken Jaw (General disorders) | 1 (1) | 1 (1)
Difficulty Sleeping (Nervous system disorders) | 6 (6) | 4 (4)
Fatigue (Nervous system disorders) | 1 (1) | 4 (4)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Seizure - no loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) — Patient with history of seizure
Restless legs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Side effects of Lexapro (Psychiatric disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Assault (Social circumstances) | 0 (0) | 1 (1)
GI virus, upset, Diarrhea, gas (Gastrointestinal disorders) | 10 (11) | 4 (4)
Smashed Finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle pain/feeling achy (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
Skin Peeling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2)
Depression, increased depressive thoughts and feelings (Psychiatric disorders) | 0 (0) | 3 (3)
Urinary symptoms - frequency (Renal and urinary disorders) | 1 (1) | 1 (1)
Cholecystitis (Surgical and medical procedures) | 1 (1) | 0 (0)
Poor concentration (Psychiatric disorders) | 0 (0) | 2 (2)
Decreased energy (Psychiatric disorders) | 0 (0) | 2 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (2)
Increased score in suicidal thoughts question (Psychiatric disorders) | 4 (4) | 2 (2) — Patient Health Questionnaire-9 (PHQ-9) individual score of suicidal thoughts question was non-zero from previous assessments.
Fainting during blood draw (General disorders) | 2 (2) | 0 (0)
Dry Mouth (General disorders) | 2 (2) | 1 (1)
Edema/bloating after starting meds & increased on full dose (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Gabapentin started same day as study med
Altered mental status due to hepatic encephalopathy w/o coma (Psychiatric disorders) | 1 (1) | 0 (0)
Skin Itchiness (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Relapse - alcohol consumption (Psychiatric disorders) | 4 (5) | 4 (5) — Reported from subjects who remained engaged in study participation.
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0)
Red Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Face swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pulled Hamstring (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Piercing infection (Infections and infestations) | 0 (0) | 1 (1)
Constipation (Renal and urinary disorders) | 1 (1) | 0 (0)
Possible Acamprosate side effects (Product Issues) | 1 (1) | 0 (0) — sensitive gums, nausea, headache, too hot or too cold, loss of appetite, inflammation in the knee, overall tiredness
ED visit for tooth pain (General disorders) | 1 (1) | 0 (0)
Demyelination (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — More than likely it's MS not sure at this time
Pt found unconscious & unresponsive 40-45 minutes after blood draw (Nervous system disorders) | 0 (0) | 1 (1) — consciousness returned and had 30 min of observation
Distress from symptoms with request that study psychiatrist contact them (Psychiatric disorders) | 2 (2) | 1 (1)
Shoulder injury/pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chronic Knee injury (history of) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Requires surgery after discharge
Emotional upset (Psychiatric disorders) | 2 (2) | 0 (0) — Triggered by reviewing drinking history details and marijuana use questions from the PRISM & TLFB assessments
COVID 19 (Infections and infestations) | 0 (0) | 1 (1)
Patient Health Information (PHI) shared with non-study member (Social circumstances) | 1 (1) | 0 (0) — Email w/PHI sent to HBFF employee not IRB approved - notified employee & had it deleted before opening
Mouth injury and spitting blood (General disorders) | 0 (0) | 1 (1)
Irritation, feelings of crabbiness (Psychiatric disorders) | 0 (0) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ankle injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Requires surgery
Bruise around left eye (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Panic attack with disassociation (Psychiatric disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Inpatient treatment centers were closed for a period of time and subsequently admission numbers were decreased to accommodate social distancing requirements during the COVID pandemic leading to lower recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT03818191/Prot_SAP_000.pdf